CLINICAL TRIAL: NCT03387995
Title: Safety and Efficacy of Stent Deployment for Intracranial Aneurysms: Trials of Clinical Curative Effect, Follow-up Study and Hemodynamics
Brief Title: Safety and Efficacy of Stent Deployment for Intracranial Aneurysms (SESIA)
Acronym: SESIA
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Guangdong Provincial People's Hospital (Other); Beijing Tiantan Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Affiliated Hospital Of Southwest Medical University (Other); Guangdong 999 Brain Hospital (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Duan Chuanzhi, Neurovascular Center of Zhujiang Hospital, Zhujiang Hospital
Other Study IDs: LC2016ZD024
Record Dates: First submitted 2017-11-27; First posted 2018-01-02 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Treatment Outcome by Stent-assisted Embolization
Keywords: treatment outcome
MeSH Terms: interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Anterior communicating artery aneurysm: Contains 5 subgroups: LVIS stent, Solitire stent, Enterprise stent, Neuroform stent and flow diveter stent.
  Interventions: Device: LVIS stent; Device: Solitaire stent; Device: Enterprise stent; Device: Neuroform stent; Device: Flow diverter (FD) stent
- Middle cerebral artery aneurysm: Contains 5 subgroups: LVIS stent, Solitire stent, Enterprise stent, Neuroform stent and flow diveter stent.
  Interventions: Device: LVIS stent; Device: Solitaire stent; Device: Enterprise stent; Device: Neuroform stent; Device: Flow diverter (FD) stent
- Posterior communicating artery aneurysm: Contains 5 subgroups: LVIS stent, Solitire stent, Enterprise stent, Neuroform stent and flow diveter stent.
  Interventions: Device: LVIS stent; Device: Solitaire stent; Device: Enterprise stent; Device: Neuroform stent; Device: Flow diverter (FD) stent
- Internal carotid artery aneurysm: Contains 5 subgroups: LVIS stent, Solitire stent, Enterprise stent, Neuroform stent and flow diveter stent.
  Interventions: Device: LVIS stent; Device: Solitaire stent; Device: Enterprise stent; Device: Neuroform stent; Device: Flow diverter (FD) stent
- Vertebrobasilar system aneurysms: Contains 5 subgroups: LVIS stent, Solitire stent, Enterprise stent, Neuroform stent and flow diveter stent.
  Interventions: Device: LVIS stent; Device: Solitaire stent; Device: Enterprise stent; Device: Neuroform stent; Device: Flow diverter (FD) stent

INTERVENTIONS:
Device: LVIS stent — The paitents treated by LVIS stent implantation.
Device: Solitaire stent — The paitents treated by Solitaire stent implantation.
Device: Enterprise stent — The paitents treated by Enterprise stent implantation.
Device: Neuroform stent — The paitents treated by Neuroform stent implantation.
Device: Flow diverter (FD) stent — The paitents treated by Enterprise FD implantation.

SUMMARY:
Intracranial aneurysms (IA) regarded the third cause of cerebral vascular disease is the majoy cause of subarachnoid hemorrhage (SAH). The mortality and morbidity account for 22% to 25% in cerebrovascular disease. More than half of the ruptured IA survivors has serious nerve dysfunction such as hemiplegia, aphasia,which seriously harms to human health. Endovascular embolization is one of the main treatment ways of IA.However,there are no studies on the multicenter cases of stent selection strategy at home and abroad.Therefore, the investigators conduct a prospective study by comparing the clinical efficacy, follow-up results, and hemodynamics between preoperative and postoperative patients with different types of stent assisted embolization treatment of IA.The investigators also study the relationship between cyclin dependent kinase inhibitor 2B antisense RNA 1 gene（CDKN2BAS1 gene）of IA patients and the results, for making indication of stents, improving the cure rate, reducing the recurrence rate of IA patients, providing theory gist for interventional therapy of complex IA and simplying slection of stent.

DETAILED DESCRIPTION:
Studies showed 3.6% - 6% for the incidence and 1% - 2% for the ruptctued rate of IA.The mortality and morbidity account for 22% to 25% in cerebrovascular disease ,which is a growing trend. IA is one of the major diseases which relate with people's living standards. Endovascular embolization is one of the main treatments of IA with less invasive, Better cure rates and higher safety. It has been developed rapidly and improve quality of patients' lives after treatmen.With the rapid development of neural intervention and the proliferation of specialized stents in IA, stent-assisted embolization technique is becoming more and more common .Especially, stents play an important role in intracranial aneurysmal aneurysm.

There are many kinds intracranial stents for clinical surgery, but how to choose the appropriate stent type is one of the key issues that clinicians need to settle. And, there is no relevant multicenter cases study about selection strategy of intracranial stent at home and abroad.

ELIGIBILITY:
Inclusion Criteria:

* Subject has intracranial aneurysms confirmed by CT arteriography (CTA) or magnetic resonance angiography (MRA) or digital subtraction angiography(DSA)
* Subject has accepted stent - assisted embolization or flow-diversion treatment of intracranial aneurysm

Exclusion Criteria:

* Subject has secondary intracranial aneurysms(e.g.traumatic aneurysm, infected aneurysm)
* Subject has received previous surgical clipping or endovascular treatment
* Subject has no intracranial aneurysms by DSA
* Subject with poor image quality
* Subject cannot use stent because of the small parent artery
* Subject do not need to use stent because of narrow-neck aneurysm
* History of aneurysm

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject has intracranial aneurysms confirmed by CT arteriography (CTA) or magnetic resonance angiography (MRA) or digital subtraction angiography (DSA).
Sampling Method: Non-Probability Sample
Enrollment: 4157 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
The safety evaluation of interventional therapy | 6 months later after operation
  Modified Rankin Scale (mRS) score to measure the safety of of interventional therapy
The efficacy evaluation of interventional treatment | 6 months later after operation
  Raymond-Ray scale (for common stent) and O'Kelley Morrota scale (for FD) to measure the effectiveness of interventional treatment
Evaluate the relationship between intracranial aneurysm and cyclin dependent | 6 months later after operation
  The investigators will take the participant's blood and the relationship between intracranial aneurysm and CDKN2BAS1 will be evaluated by ligase detection reaction-polymerase chain reaction(LDP-PCR)
The cerebrovascular complication after interventional therapy | 6 months later after operation
  Perioperative and delayed cerebrovascular complication after stent deployment
The incidence of in-stent stenosis after stent deployment | 6 months later after operation
  the rate and degree of in-stent stenosis after stent deployment

OTHER OUTCOMES:
The safety evaluation of interventional therapy | 24 months later after operation
  Modified Rankin Scale (mRS) score to measure the safety of of interventional therapy
The efficacy evaluation of interventional treatment | 24 months later after operation
  Raymond-Ray scale (for common stent) and O'Kelley Morrota scale (for FD) to measure the effectiveness of interventional treatment
The cerebrovascular complication after interventional therapy | 24 months later after operation
  Delayed cerebrovascular complication during follow-up
The incidence of in-stent stenosis after stent deployment | 24 months later after operation
  the rate and degree of in-stent stenosis after stent deployment

CONTACTS AND LOCATIONS:
Overall Officials: Chuanzhi Duan, Ph.D., Principal Investigator — Department of Neurosurgery, Zhujiang Hospital,Southern Medical University
Locations (1):
- ZhuJiang Hospital,Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Anonymized data that support the findings of this article can be provided upon reasonable request by the SESIA steering committee.

REFERENCES:
- [Background] Zhang X, Long XA, Luo B, Karuna T, Duan CZ. Factors responsible for poor outcome after intraprocedural rerupture of ruptured intracranial aneurysms: identification of risk factors, prevention and management on 18 cases. Eur J Radiol. 2012 Jan;81(1):e77-85. doi: 10.1016/j.ejrad.2011.02.015. Epub 2011 Feb 24. PMID 21353424
- [Background] Standhardt H, Boecher-Schwarz H, Gruber A, Benesch T, Knosp E, Bavinzski G. Endovascular treatment of unruptured intracranial aneurysms with Guglielmi detachable coils: short- and long-term results of a single-centre series. Stroke. 2008 Mar;39(3):899-904. doi: 10.1161/STROKEAHA.107.496372. Epub 2008 Feb 7. PMID 18258836
- [Background] Ishibashi T, Murayama Y, Urashima M, Saguchi T, Ebara M, Arakawa H, Irie K, Takao H, Abe T. Unruptured intracranial aneurysms: incidence of rupture and risk factors. Stroke. 2009 Jan;40(1):313-6. doi: 10.1161/STROKEAHA.108.521674. Epub 2008 Oct 9. PMID 18845802
- [Background] Gu DQ, Zhang X, Luo B, Long XA, Duan CZ. The effect of Neuroform stent-assisted coil embolization of wide-necked intracranial aneurysms and clinical factors on progressive aneurysm occlusion on angiographic follow-up. J Clin Neurosci. 2013 Feb;20(2):244-7. doi: 10.1016/j.jocn.2012.01.053. Epub 2012 Nov 30. PMID 23201094
- [Background] Ye HW, Liu YQ, Wang QJ, Zheng T, Cui XB, Gao YY, Lai LF, Zhang X, Li XF, Su SX, He XY, Duan CZ. Comparison between Solitaire AB and Enterprise stent-assisted coiling for intracranial aneurysms. Exp Ther Med. 2015 Jul;10(1):145-153. doi: 10.3892/etm.2015.2481. Epub 2015 May 8. PMID 26170926
- [Background] Li H, He XY, Li XF, Zhang X, Liu YC, Duan CZ. Treatment of giant/large internal carotid aneurysms: parent artery occlusion or stent-assisted coiling. Int J Neurosci. 2016;126(1):46-52. doi: 10.3109/00207454.2014.992427. Epub 2015 Jan 7. PMID 25565057
- [Background] Naggara ON, White PM, Guilbert F, Roy D, Weill A, Raymond J. Endovascular treatment of intracranial unruptured aneurysms: systematic review and meta-analysis of the literature on safety and efficacy. Radiology. 2010 Sep;256(3):887-97. doi: 10.1148/radiol.10091982. Epub 2010 Jul 15. PMID 20634431
- [Background] Mitra D, Herwadkar A, Soh C, Gholkar A. Follow-up of intracranial aneurysms treated with matrix detachable coils: a single-center experience. AJNR Am J Neuroradiol. 2007 Feb;28(2):362-7. PMID 17297013
- [Background] Lopes D, Sani S. Histological postmortem study of an internal carotid artery aneurysm treated with the Neuroform stent. Neurosurgery. 2005 Feb;56(2):E416; discussion E416. doi: 10.1227/01.neu.0000147977.07736.66. PMID 15670395
- [Derived] Feng X, Huang C, Tong X, Wen Z, Zhu Y, Huang M, Lin J, Huang J, Yuan H, Xu A, Ma G, Ge R, Li C, Peng C, Su S, Zhang X, Li X, Guo Z, Liu A, Duan C. Effect of LDL-Cholesterol Levels and Oral Atorvastatin on Outcomes After Pipeline Therapy for Intracranial Aneurysms. Stroke. 2025 Oct;56(10):3002-3013. doi: 10.1161/STROKEAHA.124.049833. Epub 2025 Aug 6. PMID 40765506